CLINICAL TRIAL: NCT00325910
Title: Patients With Heart Failure ANd Type 2 Diabetes Treated With Placebo Or Metformin (PHANTOM) Pilot Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient study participants
Sponsor: University of Alberta (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Approval J-2865; Ethics 6002
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure, Congestive
Keywords: Diabetes; Heart Failure; Mortality; Hospitalization; Feasability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Diabetes Mellitus | interventions — Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
To conduct a pilot study to evaluate the feasibility of a large randomized controlled trial (RCT) of metformin in patients with heart failure and type 2 diabetes and to generate initial morbidity and mortality estimates in this patient population. The primary hypothesis is that subjects with heart failure and type 2 diabetes who receive metformin will have a significant reduction in the combined endpoint of all-cause mortality and all-cause hospitalization as compared to subjects who receive placebo therapy.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a common complication of type 2 diabetes mellitus. There are limited treatment options for patients with HF and diabetes. Although metformin is considered a safe and effective medication, it is currently not recommended in patients who have HF due to a perceived increased risk of lactic acidosis. There is increasing evidence to suggest that HF does not predispose patients to increased risk of metformin induced lactic acidosis. Moreover, recent observational research has shown that metformin may be associated with reduced morbidity and mortality in diabetic HF patients as compared to sulfonylurea therapy.

Study Purpose: To conduct a pilot study to evaluate the feasibility of a large randomized controlled trial (RCT) of metformin in patients with heart failure and type 2 diabetes and to generate initial morbidity and mortality estimates in this patient population.

Study Design: A multi-centre prospective triple blinded randomized placebo controlled trial (RCT) design. Subjects will be recruited through specialist clinics (e.g., heart failure clinics, diabetes clinics), inpatient hospital admissions/emergency room visits and physician referrals in the Capital Health Region.

Subjects: All subjects with physician-diagnosed symptomatic heart failure (NYHA class I, II, III, IV) and type 2 diabetes are eligible for the study. All subjects with the following conditions will be excluded from the study: subjects currently receiving greater than 1500 mg of metformin therapy per day; subjects who are unwilling to change their antidiabetic regimens; subjects receiving insulin therapy; serum creatinine ≥ 180 μmol/L; A1c < 7.0 percent; inability to communicate (language barrier); dementia/mental illness; age < 18 years; subjects unwilling to complete self monitoring of serum blood sugars during the trial period; those participating in another heart failure or diabetes clinical trial involving medications; severe comorbidities or foreshortened life expectancy; subjects who do not provide written informed consent to participate.

Research Plan: Approximately 100 subjects will be randomly assigned to either metformin or placebo therapy. It is anticipated that enrollment for this pilot study could be accomplished within 12 months. Subjects will be prospectively followed for 6 months in duration as part of the pilot study. At time of hospital discharge or initial clinic visit, subjects will be provided with an educational package on heart failure and type 2 diabetes. They will also be provided with a medication Dosette to help maintain compliance to their medications and a clinical event diary to record clinical events in the community setting. To avoid medication intolerance, the dose of the study medication will be titrated slowly over a 2 week period in the community. Research coordinators will contact subjects weekly for the first 2 weeks to recommend dosage titration if warranted. All subjects will complete a six minute walk at both baseline at the final 6 month follow-up visits. Throughout the study, subjects will be contacted at monthly intervals for assessment of clinical endpoints. Subjects will return to the heart function clinic at 3 and 6 months for clinical assessment and to complete laboratory blood work. In addition, health related quality of life measures (i.e., EQ5D, KCCQ, RAND12) will also be collected at both baseline and the 6 month final follow-up visit.

Study outcomes: The primary outcome of the study will be a combined endpoint of all-cause mortality and all cause-hospitalization. Secondary endpoints include the individualized components of the primary outcome, development of lactic acidosis requiring urgent medical attention, change in A1c, change in six minute walk, and change in health related quality of life measures.

Data Analysis: As a pilot/feasibility stuy, a sample size of 100 patients was selected. An a priori probability of committing a type 1 error (i.e., alpha level) of 0.05 will be applied for all tests of statistical significance. All analyses will be conducted from an intention to treat perspective. Invesigators, patients, and data analyst will be blinded to treatment assignment. The primary outcome (all-cause mortality and hospitalization), secondary outcomes for the individual components, and risk of the development of lactic acidosis will be assessed using relative risk (RR) calculations. Secondary outcomes of change in A1c values, six minute walk, and health related quality of life from baseline to 6 months will be assessed using analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with physician-diagnosed symptomatic heart failure (NYHA class I, II, III, IV) and type 2 diabetes.

A diagnosis of type 2 diabetes defined as:

* a previous physician diagnosis of type 2 diabetes as documented in the subject's clinical record or;
* receiving oral antihyperglycemic agents or;
* a new diagnosis of type 2 diabetes during the visit within the heart failure clinic or hospital based on a fasting blood glucose ≥7.0 mmol/L or random blood glucose ≥11.1 mmol/L accompanied by acute metabolic decompensation or 2 hour plasma glucose in a 75 gram oral glucose tolerance test ≥11.1 mmol/L.

Exclusion Criteria:

* subjects currently receiving greater than 1500 mg of metformin therapy per day
* subjects who are unwilling to change their antidiabetic regimens;
* subjects receiving insulin therapy;
* serum creatinine ≥ 180 μmol/L;
* A1c < 7.0 percent;
* inability to communicate (language barrier);
* dementia/mental illness;
* age < 18 years;
* subjects unwilling to complete self-monitoring of serum blood sugars during the trial period.
* those participating in another heart failure or diabetes clinical trial involving medication;
* severe comorbidities or foreshortened life expectancy;
* subjects who do not provide written informed consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of all cause mortality and all cause hospitalization at 6 months

SECONDARY OUTCOMES:
Individual components of the primary outcome (ie death or hospitalization)
Change in A1c
Change in 6 minute walk
Change in Health Related Quality of Life
Development of Lactic Acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Johnson, PhD, Principal Investigator — University Of Alberta, Alberta, Canada
Locations (2):
- Canada (2):
  - Misericordia Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

REFERENCES:
- [Background] Eurich DT, Majumdar SR, McAlister FA, Tsuyuki RT, Johnson JA. Improved clinical outcomes associated with metformin in patients with diabetes and heart failure. Diabetes Care. 2005 Oct;28(10):2345-51. doi: 10.2337/diacare.28.10.2345. PMID 16186261
- [Derived] Eurich DT, Tsuyuki RT, Majumdar SR, McAlister FA, Lewanczuk R, Shibata MC, Johnson JA. Metformin treatment in diabetes and heart failure: when academic equipoise meets clinical reality. Trials. 2009 Feb 9;10:12. doi: 10.1186/1745-6215-10-12. PMID 19203392